CLINICAL TRIAL: NCT01597011
Title: Long-term Follow-up After Laparoscopic Inguinal Hernia Repair Using Tisseel for Mesh Fixation
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Andreas Qwist Fenger, BSc.Med., Herlev Hospital
Other Study IDs: BS12-000733
Record Dates: First submitted 2012-05-09; First posted 2012-05-11 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Hernia, Inguinal; Recurrence; Chronic Pain
Keywords: Hernia, Inguinal; Hernia repair; Fibrin Tissue Adhesive; Tisseel; Tissucol; Recurrence; Chronic Pain; Dysejaculation
MeSH Terms: conditions — Hernia, Inguinal; Recurrence; Chronic Pain | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fibrin sealant group: Patients who have undergone laparoscopic inguinal hernia repair with fibrin sealant for mesh fixation
  Interventions: Procedure: Fibrin Sealant
- Tissue-penetrating fixation group: Patients who have undergone laparoscopic inguinal hernia repair with the use of tacks, staples or sutures for mesh fixation
  Interventions: Procedure: Tissue-penetrating mesh-fixation

INTERVENTIONS:
Procedure: Fibrin Sealant — Use of fibrin sealant for mesh fixation in laparoscopic inguinal hernia repair,
  Other Names: Tisseel; Fibrin glue
  Groups: Fibrin sealant group
Procedure: Tissue-penetrating mesh-fixation — Use of tacks, staples or sutures for mesh fixation in inguinal hernia repair
  Other Names: Protacks; Hernia stapler
  Groups: Tissue-penetrating fixation group

SUMMARY:
In hernia repair a mesh is used to close the defect in the abdominal wall. This mesh is either secured with tissue penetrating devices (ex. staples,tacks or sutures) or fibrin glue (Tisseel/Tissucol) or left unfixated.

The investigators believe, and previous studies indicate, that the use of fibrin glue greatly reduces the amount of postoperative complications (ex. chronic pain, impaired ejaculation in men or recurrence of the hernia)when compared with the use of tacks or staples.

The aim of this study is to compare the recurrence rates and amount of postoperative complications in patients who have had inguinal hernia repair with fibrin glue and in patients who have had inguinal hernia repair with tacks, staples or sutures.

DETAILED DESCRIPTION:
The study will use prospectively collected data from the Danish Hernia Database to find the patients. The patients will be contacted using a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

inguinal hernia repair from January 2009-September 2012

Exclusion Criteria:

Patients lost to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled based on their registration in the Danish Hernia Database. All patients in the database who have undergone laparoscopic inguinal hernia repair from January 2009 to September 2012 will be included.
Sampling Method: Non-Probability Sample
Enrollment: 2340 (Actual)
Dates: Start 2012-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Chronic pain | within period from one year after procedure until follow-up
  Reported pain (questionnaire) from one year after procedure

SECONDARY OUTCOMES:
Recurrence | within period from procedure to follow-up
  Reherniation at repaired site. Defined as a clinically observable hernia or reoperation prior to follow-up
dysejaculation | Debut within period from procedure to follow-up
  Reported ejaculatory dysfunction in male patients

CONTACTS AND LOCATIONS:
Overall Officials: Neel M Helvind, Researcher, Principal Investigator — Herlev Hospital; Jacob Rosenberg, professor, Study Chair — Herlev Hospital; Andreas Q Fenger, Researcher, Principal Investigator — Herlev Hospital
Locations (1):
- Herlev Hospital, Herlev, Denmark